CLINICAL TRIAL: NCT00003641
Title: Phase III Randomized Study of Four Weeks of High Dose Interferon Alfa-2b in Stage T2bN0, T3a-bN0, T4a-bN0, and T1-4, N1a,2a (Microscopic) Melanoma
Brief Title: High-Dose Interferon Alfa in Treating Patients With Stage II or Stage III Melanoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); Cancer and Leukemia Group B (Network); NCIC Clinical Trials Group (Network); Children's Oncology Group (Network)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E1697; E1697 (Other: ECOG-ACRIN Cancer Research Group); U10CA023318 (NIH); CDR0000066727 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon alpha-2; Interferon-alpha; Introns; Observation; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (Other): Patients undergo observation for 4 weeks.
  Interventions: Other: observation
- Interferon Alfa-2b (Experimental): Patients receive high-dose interferon alfa-2b IV over 20 minutes daily for 5 consecutive days. Treatment repeats weekly for 4 weeks in the absence of unacceptable toxicity.
  Interventions: Biological: interferon alfa-2b

INTERVENTIONS:
Biological: interferon alfa-2b — Given IV
  Other Names: recombinant interferon alfa; Intron-A; IFN-α 2b; NSC # 377523
  Arms: Interferon Alfa-2b
Other: observation — Patients undergo observation for 4 weeks.
  Other Names: clinical observation
  Arms: Observation

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. It is not yet known whether treatment with interferon alfa is more effective than observation alone for stage II or stage III melanoma that has been completely removed surgically.

PURPOSE: This randomized phase III trial is studying high dose interferon alfa to see how well it works compared to observation only in treating patients with stage II or stage III melanoma that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

* Compare the effect of high-dose interferon alfa-2b treatment on the relapse-free survival of patients with stage II or III resected malignant melanoma.

Secondary Objectives:

* Compare the effect of this treatment regimen on overall survival of these patients.
* Assess the toxicity of this treatment in these patients.
* Compare the effect of treatment on quality of life.

OUTLINE: This is a randomized study. Patients are stratified by pathologic lymph node status (known vs unknown),lymph node staging procedures(sentinel lymph node procedure vs. elective lymph node dissection vs. no lymphadenectomy), Breslow depth (<= 1.0 mm vs. 1.01-2.0 mm vs. 2.01-4.0 mm vs > 4.0 mm), ulceration of the primary lesion (yes vs. no vs. unknown), and disease stage (lymph node positive [N1, N2a] vs. lymph node negative [N0]). Patients are randomized into one of two treatment arms in a 1:1 ratio.

* Arm I (observation): Patients undergo observation for 4 weeks.
* Arm II (Interferon Alfa-2b): Patients receive high-dose interferon alfa-2b intravenously (IV) over 20 minutes daily for 5 consecutive days. Treatment repeats weekly for 4 weeks in the absence of unacceptable toxicity.

Quality of life is assessed before treatment, at day 22, every 3 months for 2 years, and then every 6 months for 3 years.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter until 15 years after randomization.

PROJECTED ACCRUAL: A total of 1,420 patients will be accrued for this study over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary melanoma of cutaneous origin

  * Stage II (T3 N0 M0 1.5-4.0 mm Breslow depth)

    * Clinically negative regional lymph node pathologic status unknown OR
    * Histologically negative regional lymph nodes
  * Stage III (T4 N0 M0)

    * Greater than 4.0 mm Breslow depth OR
  * Stage III (T1-4 N1)

    * One lymph node positive microscopically
* Patients must meet at least 1 of the following criteria:

  * T2b N0 - primary melanoma 1.01-2.0 mm with ulceration, node negative
  * T3a-b N0 - primary melanoma 2.01-4.0 mm with and without ulceration, node negative
  * T4a-b N0 - primary melanoma > 4.0 mm with or without ulceration, node negative
  * T1a N1a-2a (microscopic) - primary melanoma of any thickness with microscopically positive lymph node (any number)
* Patients with a positive sentinel node should undergo complete lymphadenectomy of the nodal basin prior to study
* Must complete all primary therapy (wide excision with or without lymphadenectomy) and be randomized in this study within 84 days of wide excision
* Must have undergone an adequate wide excision of the primary lesion
* Age 18 and over (For ECOG patients only, patients must be >=10 years)
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1
* Adequate hematopoietic, hepatic, and renal function based on the following tests:

  * White blood cell (WBC) cout at least 3,000/mm^3
  * Platelet count at least 125,000/mm^3
  * Hematocrit at least 30%
  * Bilirubin no greater than 2 times upper limit of normal (ULN)
  * Aspartate aminotransferase (AST), lactate dehydrogenase (LDH), and alkaline phosphatase no greater than 2 times ULN
  * If lactate dehydrogenase or alkaline phosphatase is above normal, a contrast-enhanced computed tomography (CT) scan or Magnetic resonance imaging (MRI) of the liver is required to document the absence of tumor
  * Blood urea nitrogen (BUN) no greater than 33 mg/dL OR Creatinine no greater than 1.8 mg/dL
* No other concurrent or prior malignancies within the past 5 years except:

  * Cancer in situ
  * Lobular carcinoma in situ of the breast
  * Carcinoma in situ of the cervix
  * Atypical melanocytic hyperplasia or Clark 1 melanoma in situ
  * Basal or squamous cell skin cancer
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study

Exclusion Criteria:

* Clinical, radiological/laboratory, or pathological evidence of incompletely resected melanoma or any distant metastatic disease
* Clinically palpable lymphadenopathy
* Evidence of organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that would preclude study participation
* Other significant medical or surgical condition, or any medication or treatment regimens, that would interfere with study participation
* Pregnant or nursing
* Other history of invasive melanoma
* Autoimmune disorders or conditions of immunosuppression
* History of active ischemic heart disease
* Cerebrovascular disease
* Congestive heart failure (New York Heart Association class III or IV heart disease)
* Prior or concurrent chemotherapy
* Prior immunotherapy including tumor vaccines, interferon, interleukins, levamisole, or other biologic response modifiers for melanoma
* Concurrent systemic corticosteroids including oral steroids (i.e., prednisone, dexamethasone), topical steroid creams or ointments, or any steroid-containing inhalers
* Prior or concurrent radiotherapy
* Other concurrent immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 1999-03-25 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv S. Agarwala, MD, Study Chair — St. Luke's Cancer Network at St. Luke's Hospital; John M. Kirkwood, MD, Study Chair — UPMC Cancer Center at UPMC Presbyterian; Lawrence E. Flaherty, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; William E. Carson, MD, Study Chair — Ohio State University Comprehensive Cancer Center; Michael Smylie, MD, MB, ChB, Study Chair — Cross Cancer Institute at University of Alberta; Alberto S. Pappo, MD, Principal Investigator — Texas Children's Cancer Center
Locations (533):
- United States (511):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente - Deer Valley, Antioch, California
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Southern California Permanente Medical Group, Downey, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Sutter Health - Western Division Cancer Research Group, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Kaiser Permanente - Denver, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Kaiser Permanente - Lafayette, Lafayette, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Carl and Dorothy Bennett Cancer Center at Stamford Hospital, Stamford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Kaiser Permanente - Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Hematology Oncology Associates of Illinois - Berwyn, Berwyn, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Saint Joseph Hospital, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Evanston Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - La Grange Oncology Associates - Geneva, Naperville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Michiana Hematology Oncology PC - La Porte, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Medical Consultants, PC at Ball Memorial Cancer Center, Muncie, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Care at Our Lady of Bellefonte Hospital, Ashland, Kentucky
  - Drs. Carrol, Sheth, Raghavan, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Michiana Hematology Oncology PC - Niles, Niles, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls Medical Group, PA, Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center at Catholic Medical Center, Manchester, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Susquehanna Cancer Center at Divine Providence Hospital, Williamsport, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Center for Biomedical Research, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Harrison Poulsbo Hematology and Onocology, Poulsbo, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology, PS, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Schiffler Cancer Center at Wheeling Hospital, Wheeling, West Virginia
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Aurora Memorial Hospital of Burlington, Burlington, Wisconsin
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Oncology Alliance - Franklin, Franklin, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Vince Lombardi Cancer Clinic - Green Bay at Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Oncology Alliance - Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic - Marinette, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Advanced Healthcare East Mequon Clinic, Mequon, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Oncology Alliance, SC - Milwaukee - South, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Aurora Health Center - Racine, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Aurora Health Center - Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Oncology Alliance, SC - Milwaukee - West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales, Australia
- Canada (20):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Royal Victoria Hospital of Barrie, Barrie, Ontario
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - R. S. McLaughlin Durham Regional Cancer Centre at Lakeridge Health Oshawa, Oshawa, Ontario
  - St. Catharines General Hospital at Niagara Health System, St. Catharines, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Trillium Health Centre - Mississauga Site, Toronto, Ontario
  - Windsor Regional Cancer Centre at Windsor Regional Hospital, Windsor, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
- Pretoria Academic Hospital, Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on December 22, 1998, accrued its first patient on March 25, 1999, and closed to accrual on October 26, 2010 with final accrual of 1150 patients
Period: Overall Study
Arm/Group | Observation | Interferon Alfa-2b
Started | 569 | 581
Treated | 2 (Patients on arm I should undergo observation, but 2 patients received interferon therapy) | 569
Toxicity Assessed | 439 (439 patients on arm I had their toxicity assessed even though they did not receive any treatment) | 568
Completed | 0 | 407
Not Completed | 569 | 174
Not completed — Withdrawal by Subject | 0 | 100
Not completed — Adverse Event | 0 | 38
Not completed — Disease progression | 0 | 2
Not completed — Unknown/missing | 0 | 22
Not completed — Should not receive interferon therapy | 2 | 0
Not completed — Never started interferon | 567 | 12

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Interferon Alfa-2b | Total
Number analyzed (Participants) | 569 | 581 | 1150
Age, Continuous [Median (Full Range); unit: years] | 52 [19 to 81] | 52 [10 to 85] | 52 [10 to 85]
Sex/Gender, Customized [Number; unit: participants] — 1 patient on arm I and 1 patient on arm II had missing information about sex
  participants
    Female | 248 | 244 | 492
    Male | 320 | 336 | 656
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: 5-year Relapse-free Survival Rate
Description: Relapse-free survival (RFS) was defined as time from randomization to disease relapse or death from any cause, whichever occurred first. Patients without disease relapse were censored at last disease assessment date known of free of relapse. Kaplan-Meier method was used to estimate 5-year RFS rate in the intent-to-treat (ITT) patients.
Time Frame: assessed every 3 months for 2 years, every 6 months for 3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Observation | Interferon Alfa-2b
Number analyzed (Participants) | 569 | 581
proportion of participants | 0.70 [0.66 to 0.74] | 0.70 [0.66 to 0.74]
Statistical Analysis 1: Comparison: Observation vs Interferon Alfa-2b; Test type: Superiority or Other; p = 0.964, Log Rank; stratified on the stratification factors used for randomization

2. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival (OS) was defined as time from randomization to death from any cause. Patients still alive were censored at last known alive date. Kaplan-Meier method was used to estimate 5-year OS rate in the ITT patients.
Time Frame: assessed every 3 months for 2 years, every 6 months for 3 years
Population: all randomized patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Observation | Interferon Alfa-2b
Number analyzed (Participants) | 569 | 581
proportion of participants | 0.83 [0.79 to 0.86] | 0.83 [0.80 to 0.86]
Statistical Analysis 1: Comparison: Observation vs Interferon Alfa-2b; Test type: Superiority or Other; p = 0.558, Log Rank; Stratified on the stratification factors used for randomization

ADVERSE EVENTS:
Time Frame: Assessed at the end of treatment (4 weeks) and for 30 days following the last dose of protocol drug, or until the initiation of subsequent treatment, whichever comes first
Description: Prior to diagnosis of relapse, any severe (Grade ≥ 3) long term toxicity that has not been previously reported was collected via the long-term follow up form, assessed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter until 15 years after randomization.These long term toxicities were included here as well.
Groups:
- Interferon Alfa-2b: Patients receive high-dose interferon alfa-2b IV over 20 minutes daily for 5 consecutive days
Arm/Group | Observation | Interferon Alfa-2b
Serious Adverse Events (participants affected / at risk) | 20/439 | 325/568
Other Adverse Events (participants affected / at risk) | 74/439 | 558/568
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=439) | Interferon Alfa-2b (N=568)
Allergic reaction (Immune system disorders) | 0 | 1
INNER EAR/HEARING (Ear and labyrinth disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytes decreased (Investigations) | 0 | 38
Neutrophils decreased (Investigations) | 8 | 130
Platelets decreased (Investigations) | 0 | 3
Hematologic-other (Blood and lymphatic system disorders) | 0 | 1
Supraventricular arrhythmias (Cardiac disorders) | 0 | 1
Vasovagal episode (Nervous system disorders) | 0 | 1
Cardiac-ischemia (Cardiac disorders) | 0 | 2
Cardiac-left ventric (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 5
Hypotension (Vascular disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Thrombosis/embolism (Vascular disorders) | 0 | 1
Fatigue (General disorders) | 0 | 70
Fever (General disorders) | 0 | 4
Rigors/chills (General disorders) | 0 | 1
CONSTITUTIONAL (General disorders) | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 5
Anorexia (Metabolism and nutrition disorders) | 0 | 11
Constipation (Gastrointestinal disorders) | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 28
STOMATITIS (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 19
GI-other (Gastrointestinal disorders) | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 4
GGT increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 74
Alanine aminotransferase increased (Investigations) | 0 | 30
Catheter-related infection (Infections and infestations) | 0 | 1
Infection w/ grade 3 or 4 neutropenia (Infections and infestations) | 0 | 2
INFECTION W/ UNKNOWN ANC (Infections and infestations) | 0 | 2
Infection w/o neutropenia (Infections and infestations) | 0 | 2
INFECTION-OTHER (Infections and infestations) | 0 | 2
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 4
Depressed level of consciousness (Nervous system disorders) | 0 | 3
Dizziness/lightheadedness (Nervous system disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 5
Memory loss (Nervous system disorders) | 0 | 1
Anxiety/agitation (Psychiatric disorders) | 0 | 6
Depression (Psychiatric disorders) | 0 | 11
Neuropathy-cranial (Nervous system disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 3
Seizure (Nervous system disorders) | 0 | 1
Speech impairment (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 3
VERTIGO (Nervous system disorders) | 0 | 1
Neurologic-other (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 13
Pain-other (General disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Creatinine increased (Investigations) | 6 | 13
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=439) | Interferon Alfa-2b (N=568)
Anemia (Blood and lymphatic system disorders) | 12 | 123
Leukocytes decreased (Investigations) | 6 | 321
Neutrophils decreased (Investigations) | 4 | 283
Platelets decreased (Investigations) | 2 | 200
Fatigue (General disorders) | 11 | 454
Fever (General disorders) | 0 | 256
Rigors/chills (General disorders) | 0 | 342
Sweating (Skin and subcutaneous tissue disorders) | 0 | 83
Weight loss (Investigations) | 0 | 120
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 30
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 64
Anorexia (Metabolism and nutrition disorders) | 0 | 283
Constipation (Gastrointestinal disorders) | 2 | 106
Nausea (Gastrointestinal disorders) | 1 | 340
Taste disturbance (Nervous system disorders) | 0 | 176
Vomiting (Gastrointestinal disorders) | 0 | 133
GI-other (Gastrointestinal disorders) | 0 | 41
Alkaline phosphatase increased (Investigations) | 2 | 69
Blood bilirubin increased (Investigations) | 2 | 43
Aspartate aminotransferase increased (Investigations) | 8 | 373
Alanine aminotransferase increased (Investigations) | 4 | 80
Dizziness/lightheadedness (Nervous system disorders) | 0 | 95
Insomnia (Psychiatric disorders) | 3 | 113
Anxiety/agitation (Psychiatric disorders) | 7 | 91
Depression (Psychiatric disorders) | 4 | 90
Neuropathy-sensory (Nervous system disorders) | 8 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 137
Headache (Nervous system disorders) | 8 | 270
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 229
Pain-other (General disorders) | 17 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less